CLINICAL TRIAL: NCT03591289
Title: Does Depth of Neuromuscular Blockade (NMB) Affect Surgical Conditions and Postoperative Pain in Obese Patients Undergoing Robotic Surgery
Brief Title: Does Depth of Neuromuscular Blockade (NMB) Affect Surgical Conditions in Obese Patients Undergoing Robotic Surgery
Acronym: NMB
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: study never started up at site
Sponsor: Rainer Lenhardt (Other)
Responsible Party: Sponsor-Investigator, Rainer Lenhardt, Professor and Vice-Chair Clinical Affairs; Department of Anesthesiology and Perioperative Medicine, MBA, University of Louisville
Organization: University of Louisville (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17.1119
Record Dates: First submitted 2017-11-03; First posted 2018-07-19 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-04

CONDITIONS: GYN Disorders; Urologic Diseases
Keywords: Robotic Surgery
MeSH Terms: conditions — Genital Diseases, Female; Urologic Diseases | interventions — Rocuronium

STUDY DESIGN:
Intervention Model Description: two different regimens (doses) of two drugs (Rocuronium, Sugammadex)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Subjects will not be informed to which NMB depth they were randomized to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Deep NMB (Active Comparator): Deep NMB: Intervention: Rocuronium will be given as a continuous infusion for deep block. TOF will be maintained at 0 (zero) with at least one PTC. Patients' paralysis will be continued through the anesthesia period. At the end of surgery, patients will receive 4 mg/kg sugammadex and the patient's trachea will be extubated according to routine extubation criteria.
  Interventions: Drug: NMB with rocuronium bromide
- Moderate NMB (Active Comparator): Moderate NMB: Intervention: Rocuronium will be used as bolus doses to achieve a moderate block. TOF will be maintained between 1 to 3 twitches. PTC will not be counted. Paralysis will be continued throughout the anesthesia period. At the end of surgery, patients will receive 2 mg/kg sugammadex and the patient's trachea will be extubated according to routine extubation criteria.
  Interventions: Drug: NMB with rocuronium bromide

INTERVENTIONS:
Drug: NMB with rocuronium bromide — Moderate versus deep neuromuscular block Not a device study
  Other Names: Reversal with suggammadex

SUMMARY:
A prospective, randomized, outcome trial to evaluate, if depth of neuromuscular blockade (NMB) will affect surgical conditions and postoperative pain based on the degree of neuromuscular block during robotic surgery for gynecological and urologic procedures in obese and non-obese patients.

DETAILED DESCRIPTION:
Study Procedures:

Anesthesia will be induced with propofol (2 mg/kg), fentanyl (1-2 µg/kg) and rocuronium (0.6 mg/kg) to facilitate intubation. A #8 endotracheal tube in males and #7endotracheal tube in females will be inserted in the trachea and secured at 22 cm. Anesthesia will be maintained with sevoflurane to maintain the BIS value between 40 and 60. Analgesia will be provided with fentanyl at 1-2 µg/kg/h or remifentanil 0.5-2 µg/kg/min. Anesthesia will continue until surgery is completed.

Patients will be randomized to either deep neuromuscular blockade (NMB) or moderate NMB as described below.

Rocuronium will be administered to keep NMB deep or moderate NMB according to the randomization.

Deep NMB: Rocuronium will be given as a continuous infusion for deep block. Train of four (TOF) will be maintained at 0 (zero) with at least one post-tetanic count (PTC). Patients' paralysis will be continued through the anesthesia period. At the end of surgery, deep Block patients' will receive 4 mg/kg sugammadex and the patient's trachea will be extubated according to routine extubation criteria.

Moderate NMB: Rocuronium will be used as bolus doses to achieve a moderate block. TOF will be maintained between 1 to 3 twitches. PTC will not be counted. Paralysis will be continued throughout the anesthesia period. At the end of surgery, patients will receive 2 mg/kg sugammadex in the moderate NMB and the patient's trachea will be extubated according to routine extubation criteria.

NMB will be assessed by acceleromyography (STIMPOD NMS410 Peripheral Nerve Stimulator, Xavant Technology (Pty) Ltd. Silverton, Pretoria, South Africa)

The ventilator will be set at pressure-controlled mode and patients will be ventilated with an airway pressure corresponding to a tidal volume of 8 mL/kg up to a maximum airway pressure of 35 cmH20. Inspired oxygen will be kept near 50% but will be increased if necessary to maintain a hemoglobin oxygen saturation ≥95%. PEEP will be set at 5 cmH20. Respiratory rate will be 12 breaths per minute.

Patients' will have a small finger cuff (finger plethysmography) with a transducer and continuous real-time cardiovascular monitor (Edwards, Life Science, Irvine, CA) The patient may also receive an arterial catheter (radial artery) for continuous real-time cardiovascular monitoring based on the clinicians' preference. Arterial waveform will be recorded continuously. A pulse oximeter (LNOP Adt, Masimo Corp, Irvine, CA) will be attached to the index finger of the patient's same hand and connected to a bedside monitor (Radical 7, Masimo Corp, Irvine, CA); the oximeter will be wrapped to prevent interference from outside light. Perfusion variability index (PVI) calculates the respiratory variations in the plethysmography waveform amplitude (Perfusion index [PI]) using the maximum and minimum PI values over a given time period.

Intraoperative fluid management will be performed with normosol 2 mL/kg/h. Fluid boluses will be given as guided by stroke volume variation (SVV). Hetastarch will be given as a bolus in 250 mL increments to a maximum of 50 mL/kg. The fluid bolus will be given over 2 minutes. A bladder (foley) catheter will be inserted after induction of anesthesia. This is part of conventional care and allows for more accurate fluid volume tracking.

Once the patient is in Trendelenburg position and should a measurement yield that SVV is staying above 10%, a fluid bolus of 250 mL of hetastarch will be given over 2 minutes and repeated until the SVV falls below 10%.

During abdominal CO2 insufflation, the intra-abdominal pressure will be kept at 15 cmH2O. The Trendelenburg position will be 30º, which corresponds to the maximum inclination of the OR table.

Postoperatively, patients will receive a bilateral transverse abdominal plane (TAP) block with ropivacaine in the post-operative area. Patients will receive a PCA pump with hydromorphone for pain management.(This is all standard practice).

Measurements:

A) Measurements that will be recorded once the patient is brought into the operating room and throughout the intraoperative period include:

1. Hemodynamic data; Systolic, diastolic and mean arterial blood pressure in mmHg, Cardiac Output and Cardiac Index in liters per minute, Stroke Volume Variation in percent, Pulse Pressure Variation in percent, Perfusion Index (number from 0.1-10, no units), Perfusion Variability Index in percent

Time points the data will be recorded include:

1. After patients placement on operative table, while still awake, lying flat for one minute but prior to induction.
2. Intraoperative, one minute after induction of anesthesia and intubation
3. Intraoperative, one minute after initiation of pneumoperitoneum, with just one trocar placed
4. Intraoperative, one minute after positioning the patient in Trendelenburg position but before the surgeon begins
5. Intraoperative, every 15 minutes during the surgical procedure.
6. Intraoperative, when the surgeon states the surgery is completed.
7. Intraoperative, after surgery completed and one minute after reversal of Trendelenburg position.
8. Intraoperative, while the patient is still on the operative table, one minute after deflation of the peritoneum.
9. Intraoperative; additional measurements (as referred to above) may be recorded to capture observed changes that occurred during surgery.

B) Measurements that will be recorded after general anesthesia has been induced and throughout the intraoperative period include (same time points as above minus time point one):

2. Assessment of NMB

C) A 5-point surgical rating scale will be used to assess surgical conditions every 15 minutes:

1. The surgeon and the surgical assistant will be asked about surgical conditions every 15 minutes. Surgical conditions will be assessed by the Leiden surgical rating scale (Martini BJA 2014; 112:498).

1. Extremely poor conditions: The surgeon is unable to work due to coughing or due to the inability to obtain a visible laparoscopic field because of inadequate muscle relaxation. Additional muscle relaxants must be given.
2. Poor conditions: There is a visible laparoscopic field but the surgeon is severely hampered by inadequate muscle relaxation with continuous muscle contractions and/or movements with the hazard of tissue damage. Additional muscle relaxants must be given.
3. Acceptable conditions: There is a wide visible laparoscopic field but muscle contractions and/or movements occur regularly causing some interference with the surgeon's work. There is the need for additional muscle relaxants to prevent deterioration.
4. Good conditions: There is a wide laparoscopic working field with sporadic muscle contractions and/or movements. There is no immediate need for additional muscle relaxants unless there is the fear for deterioration.
5. Optimal conditions: There is a wide visible laparoscopic working field without any movement or contractions. There is no need for additional muscle relaxants.

2. Intraoperatively; The Intra-abdominal pressures (mmHg) will be recorded every 15 minutes during the surgery. The amount of flow and the total amount of CO2 (in liters) will be recorded.

3. Forearm - fingertip temperature gradients will be measured by Mon-a-thermometer (Mallinckrodt Medical, Inc. St. Louis, MO) and disposable Mon-a-therm thermocouples. Vasoconstriction will be identified when forearm - fingertip temperature gradient is ≥ 00 Cº and PI < 1.

D) Additional assessments:

1. Intraoperatively; the surgical assistant will report any episode(s) of abdominal contractions throughout the surgery.
2. The degree of the patients' Trendelenburg position will be measured intra-operatively with an angle ruler.
3. The amount of rocuronium received intraoperatively, during the course of surgery, will be recorded.

Subjects demographic information will be collected at the time of consent. This will include, age, gender, weight in kilograms, height in centimeters, BMI in kg/m^2, waist-to hip ratio, surgical procedure and co-morbidities.

E) Post-operative assessments:

1. Pain assessments will be completed using the "visual pain analogue scale" (VAS scale from 1 to 100 mm, with 1 meaning no pain at all to 100 rated as the worst pain imaginable). Assessments will be completed by a study team member. Patients will be asked about their pain level by visual analogue scale at the following time points:

   1. Baseline; in pre-operative holding area
   2. One hour after admission to PACU, post-operatively
   3. Six hours postoperatively
   4. Post-operative day one (next morning) between 0600 and 1000
2. Postoperative hydromorphone PCA requirement will be recorded up until the post-operative DAY ONE (Overall amount of hydromorphone measured in milligrams total). Pain assessment will be completed between 0600 and 1000 am.

All other pain management (rescue) medications the patient received up to the time of the "AM" post-operative assessment will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for elective robotic gynecological or urologic surgery under general anesthesia.
2. Patients are willing and sign an IRB approved consent
3. Patients will be 18 years or older

Exclusion Criteria:

1. Patients with atrial fibrillation
2. Other significant arrhythmia (Lown grade 3 or greater)
3. Patients with aortic regurgitation
4. Unable to receive or refuses to usehydromorphone for pain management post-operatively (allergic, bad experience previously with use)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-02 (Estimated); Primary Completion 2018-02 (Estimated); Study Completion 2018-07-12 (Actual)

PRIMARY OUTCOMES:
Assessment of surgical conditions during deep versus moderate NMB in patients undergoing robotic abdominal surgery | data will be reported every 15 minutes starting post anesthesia induction until the end of general anesthesia
  Surgical conditions will be assessed by the Leiden surgical rating scale (Martini BJA 2014; 112:498) as follows:
  Scale range from 1 to 5 with 1 describing extremely poor conditions and 5 describing optimal conditions for surgery

SECONDARY OUTCOMES:
Assessment of PVI changes to predict fluid responsiveness in robotic surgery | PVI will be measured every 15 minutes and after any fluid bolus. Fluid bolus will be given, when PVI is > 12
  PVI changes will be measured after each fluid challenge and correlated with a change in stroke volume
Incidence of good and optimal surgical conditions in obese and non-obese patients undergoing robotic abdominal surgery | Data will be reported every 15 minutes starting post anesthesia induction until the end of general anesthesia
  Surgical conditions will be assessed by the Leiden surgical rating scale and will be compared in obese patients versus non-obese patients
  Surgical conditions will be assessed by the Leiden surgical rating scale (Martini BJA 2014; 112:498) as follows:
  Scale range from 1 to 5 with 1 describing extremely poor conditions and 5 describing optimal conditions for surgery
Assessment of postoperative pain after deep versus moderate NMB in patients undergoing robotic abdominal surgery. Does depth of neuromuscular block (NMB) affect postoperative pain ? | First 24 hours postoperatively at time points 1hour, 6 hours after surgery and postoperative day one
  Postoperative pain will be measured by visual pain analogue scale and by the amount of hydromorphone used in 24 hours after surgery.
  Pain assessments will be completed using the "visual pain analogue scale" (VAS). VAS scale ranges from 1 to 100 mm, with 1 meaning no pain at all to 100 rated as the worst pain imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Cooke, RN,BSN, CCRP, Study Director — University of Louisville
Locations (1):
- University of Louisville Medical School, Department of Anesthesiology and Perioperative Medicine, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No